CLINICAL TRIAL: NCT06440551
Title: Puerto Rican Obesity Intervention for Men
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Lisa Sanchez-Johnsen, Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0048231
Record Dates: First submitted 2024-04-26; First posted 2024-06-04 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Obesity
Keywords: Diet; Physical Activity; Puerto Rican
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Eating and Physical Activity - Intervention (Experimental): Participants will attend virtual classes on increasing healthy eating, increasing physical activity, and decreasing sedentary behaviors.
  Interventions: Behavioral: TeleSalud Healthy Eating- Physical Activity/Sedentary Behavior (HE-PA/SB)
- General Health Topics - Control (Active Comparator): Participants will attend virtual classes on general health topics.
  Interventions: Behavioral: TeleSalud General Health Intervention

INTERVENTIONS:
Behavioral: TeleSalud Healthy Eating- Physical Activity/Sedentary Behavior (HE-PA/SB) — Participants will meet via telehealth for 4 months (twice a week for 3 months and then once per week for 1 month) for a TeleSalud HE-PA/SB Class, after which they will attend one maintenance meeting per month for 4 months. Weekly, Day 1 (Healthy Eating & PA-SB Class): Participants will receive a 50-min. healthy eating class. Physical Activity- Sedentary Behavior (PA-SB) Class: By discussing barriers and strategies to overcome barriers, this will help to increase self-efficacy. We will engage in Latino-centered moderate impact (increasing to vigorous) aerobics with Latino or salsa movements and music for 45-50 minutes. Aspects of kickboxing aerobics will be integrated. Goal: Exercise a minimum of 150-250 min./ week of moderate intensity. Weekly, Day 2: PA-SB identical PA-SB to Day 1. Maintenance (Months 5-8): Meetings once/ month for 70 min. for HE/PA-SB class, including 25 min. to discuss diet and PA-SB barriers. Goal: Exercise a minimum of 150-250 min./week.
  Arms: Healthy Eating and Physical Activity - Intervention
Behavioral: TeleSalud General Health Intervention — Weekly: Participants will meet via telehealth for 4 months (twice a week for 3 months and then once per week for 1 month) for a TeleSalud General Heath Class, after which they will attend one maintenance meeting per month for 4 months. Participants will meet and discuss general health topics (not diet or PA). Examples of the general health topics are: Back Pain, Muscle Strains, Alcohol Use, Stress & Coping, Oral and Dental Health, Safety Tips, Emergency Preparedness. The content is relevant to Latinos, and information is focused on Latino men. Maintenance (Months 5-8): Participants will meet via telehealth once/ month for 70 min. to discuss general health topics. To enhance motivation to complete the study and assessments, this group will receive a copy of the TeleSalud HE-PA/SB intervention manual and related materials after the maintenance period ends.
  Arms: General Health Topics - Control

SUMMARY:
The goal of this clinical trial is to address the high rates of overweight/obesity in Puerto Rican (PR) men. The main question it aims to answer is whether virtual culturally relevant classes supporting physical activity and healthy eating for Puerto Rican men at different levels of acculturation to the US culture, will help these men achieve clinically meaningful weight loss.

The purpose of this project is to assess whether a virtual intervention tailored for Puerto Rican men that includes information about healthy eating, physical activity, sedentary behavior is feasible and acceptable compared to a general health (GH) intervention. It is also to determine whether this intervention leads to healthier eating, increased physical activity, less sedentary behavior (low activity), and clinically meaningful weight loss.

Hypothesis 1: Test the feasibility (recruitment, retention, adherence, fidelity) and acceptability (treatment components, intervention leaders, telehealth modality, technology and equipment, intervention satisfaction, satisfaction with randomized study, and measures) of a randomized 4-month synchronous telehealth lifestyle intervention led by a community health promoter and behavioral health specialist, who will receive either: TeleSalud HE-PA/SB" or TeleSalud GH in 48 PR men.

Hypothesis 2: Demonstrate proof -of-concept by achieving a clinically significant weight reduction of ≥ 5% of baseline weight in the TeleSalud HE-PA/SB intervention after 4 months and at the end of the 4-month maintenance compared to the TeleSalud General Health intervention.

Researchers will compare this to a group that will receive information about general health topics - not healthy eating or physical activity.

* Participants in both groups will meet via virtually for 4 months (twice per week for 3 months and once per week for 1 month).
* Participants will then meet one per month for a maintenance session for the next 4 months.

ELIGIBILITY:
Inclusion criteria:

1. Male of Puerto Rican descent over 35 years.
2. BMI ≥25 by anthropometrically measured weight and height.
3. Physically able to exercise (via the EASY tool [106, 107]; Appendix 2). If responses to the EASY indicate that medical clearance is needed, then able to receive medical clearance to participate in the study.
4. Has access to secure computer or tablet in a private location with reliable internet connection to support video streaming
5. Ability to understand and speak English. For those without a high-speed internet and private space to exercise, we will work with our community partners to identify a space with access to videoconferencing so they can attend the telehealth class.

Exclusion:

1. Does not understand/speak English.
2. Plans to move from the Illinois area during the study.
3. Currently in a formal weight management program.
4. Current or planned use of weight control or loss medication prescribed by a doctor.
5. Currently exercising >1 time/week.
6. Unable to attend study times.
7. Serious medical problems or medications that would make protocol compliance difficult or dangerous, e.g., unable to engage in moderate & eventually vigorous exercise, uncontrolled diabetes (A1C > 9) or hypertension (systolic >160 or diastolic >100), hypoglycemia, heart attack in the past six months, unstable angina, life-threatening arrhythmias, cancer that required treatment in the last 5 years (except non-melanoma skin cancers that have been cured). Patients who have been treated for cancer in the past 5 years may require different diet and PA recommendations than individuals without treatment for cancer in the past 5 years.
8. In the EASY interview, if participant answers yes to the question that indicates they fall or always use an assisted device while walking.
9. Current alcohol abuse (>35 alcoholic drinks/week); score of yes to > 2 questions on the CAGE alcohol scale (Appendix 1) [108].

Min Age: 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-10-15 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability- Fidelity: Delivery | 4 months, 8 months
  Delivery will be measured by an adherence checklist. It will monitor consistency and accuracy in the delivery of the intervention.
Acceptability- Fidelity: Receipt | 4 months, 8 months
  Receipt will be measured by participants' self-reports of understanding and knowledge acquisition of content for both groups.
Acceptability- Fidelity: Enactment | 4 months, 8 months
  Enactment will be measured by participants' self-report of changes in behavior based on targets of treatment (e.g., Healthy Eating, Physical Activity, and Sedentary Behavior, General Health.)
Acceptability- Helpfulness of Treatment Components | 4 months, 8 months
  Perceived helpfulness/ effectiveness of various treatment components (12 questions, on a 5- point Likert scale: not at all to extremely effective) will be assessed. The average of the treatment component questions will be used as the overall dependent measure of the acceptability of the treatment components.
Acceptability- Helpfulness/ Effectiveness of the Intervention Leaders | 4 months, 8 months
  Perceived helpfulness/ effectiveness of the intervention leaders (6 questions, on a 5-point Likert scale: not at alll to extremely helpful) will be assessed. The average of the questions will be used as the overall dependent measures of the acceptability of the intervention leaders.
Acceptability- Intervention Satisfaction | 4 months, 8 months
  Acceptability- Assessed by an intervention satisfaction questionnaire (14 questions, on a 5- point Likert scale: not at all satisfied to extremely satisfied).
Acceptability- Perceived Helpfulness/ Effectiveness of the Telehealth Modality, Technology, and Equipment | Baseline, 4 months, 8 months
  Perceived helpfulness/ effectiveness of the telehealth modality, technology and equipment (3 questions, on 5-point Likert scale: not at all to extremely effective) will be assessed. The average of the telehealth components questions will be used as the overall dependent measure of the acceptability of the telehealth components.
Acceptability- Satisfaction with Random Assignment to Groups | Baseline, 4 months, 8 months
  Acceptability- Assessed by a questionnaire assessing satisfaction with being in a study with random assignment to groups (14 questions, on a 5-point Likert scale: not at all satisfied to extremely satisfied).
Dietary Intake: Number of Servings of Fruits | Baseline, 4 months, 8 months
  Changes in number of servings of fruits will be measured by the Automated Self-Administered 24- Hour (ASA24) Dietary Assessment Tool.
Dietary Intake: Number of Servings of Vegetables | Baseline, 4 months, 8 months
  Change in number of servings of vegetables will be measured by the Automated Self-Administered 24- Hour (ASA24) Dietary Assessment Tool.
Dietary Intake: Percent of Calories from Saturated Fat | Baseline, 4 months, 8 months
  Changes in percent of calories from saturated fat will be measured by the Automated Self-Administered 24-Hour (ASA24) Dietary Assessment Tool.
Dietary Intake: Total Energy Intake | Baseline, 4 months, 8 months
  Changes in total energy intake will be measured by the Automated Self-Administered 24-Hour (ASA24) Dietary Assessment Tool.
Feasibility- Adherence- Monthly Attendance | 4 months, 8 months
  Feasibility- Adherence- Monthly: Will be measured by the frequency of attendance at each session on a monthly basis.
Feasibility- Adherence- Number of Make-Up Sessions | 4 months, 8 months
  Feasibility- Adherence- Number of Make-Up Sessions: Will be assessed by frequency/counts of number of make-up sessions.
Feasibility- Adherence- Number of Missed Sessions Overall | 4 months, 8 months
  Feasibility- Adherence- Number of Missed Sessions Overall: Will be assessed by frequency/ counts of the number of missed sessions overall (no make-up sessions).
Feasibility- Adherence- Weekly Attendance | 4 months, 8 months
  Feasibility- Adherence- Weekly Attendance: Will be measured by the frequency of attendance at each session on a weekly basis.
Feasibility- Recruitment- Number Enrolled | Pre-Intervention
  Recruitment feasibility assessed by the number of participants enrolled.
Feasibility- Recruitment- Number of Contacts | Pre-Intervention
  Recruitment feasibility assessed by counts of the number of contacts.
Feasibility- Recruitment- Rate of Consenting | Pre-Intervention
  Recruitment feasibility assessed by the rate of consenting.
Feasibility- Recruitment- Rate of Enrollment | Pre-Intervention
  Recruitment feasibility assessed by the rate of enrollment.
Feasibility- Recruitment- Rate of Screening | Pre-Intervention
  Recruitment feasibility assessed by the rate of screening.
Feasibility- Recruitment- Recruitment Method | Pre-Intervention
  Feasibility assessed by tracking the method of recruitment.
Feasibility- Recruitment- Response Rate | Pre-Intervention
  Recruitment feasibility assessed by rate of response.
Feasibility- Recruitment- Type of Contact | Pre-Intervention
  Recruitment feasibility assessed by tracking the type of contact.
Feasibility- Retention- Number Completed the intervention | 4 months, 8 months
  Retention assessed by counts and frequency of the number who completed the interventions.
Feasibility- Recruitment- Number Screened | Pre-Intervention
  Recruitment feasibility assessed by the count of number of individuals screened.
Feasibility- Retention- Number of Classes Attended | 4 months, 8 months
  Retention- assessed by counts of the number of classes attended.
Feasibility- Retention- Percent Completed the Interventions | 4 months, 8 months
  Retention assessed by the percent of participants who completed the interventions.
Feasibility- Retention- Percent of Classes Attended | 4 months, 8 months
  Retention assessed by percent of classes attended.
Feasibility- Recruitment- Number Consented | Pre-Intervention
  Recruitment feasibility assessed by the number of participants who consented.
Objective Physical Activity (Accelerometer) | Baseline, 4 months, 8 months
  A triaxial wrist accelerometer (ActiGraph wGT3XBT) will measure objective physical activity. They will used the accelerometer during waking hours for 7 days on their non-dominant wrist.
Subjective Physical Activity (International Physical Activity Questionnaire) | Baseline, 4 months, 8 months
  The International Physical Activity Questionnaire long form- will measure sedentary and leisure and non-leisure time physical activity.
Subjective Sedentary Behavior (International Physical Activity Questionnaire) | Baseline, 4 months, 8 months
  The International Physical Activity Questionnaire long form- will measure sedentary and leisure and non-leisure time physical activity.

SECONDARY OUTCOMES:
Body Mass Index | Baseline, 4 months, 8 months
  Body Mass Index (BMI) will be assessed by objectively measured height and weight.
Outcome Expectations for Diet Questionnaire | Baseline, 4 months, 8 months
  Outcome expectations will be assessed by the Outcome Expectations for Diet Questionnaire. This measure will be used to assess the various components of Social Cognitive Theory which are guiding the TeleSalud HE-PA/SB intervention.
Exercise Outcomes on the Outcomes Expectations Questionnaire | Baseline, 4 months, 8 months
  Outcome expectations for Exercise will be assessed by the Exercise Outcomes on the Outcomes Expectations Questionnaire. This measure will be used to assess the various components of Social Cognitive Theory which are guiding the TeleSalud HE-PA/SB intervention.
Self-Efficacy for Dietary Behaviors | Baseline, 4 months, 8 months
  Self-efficacy will be assessed by the Self-Efficacy for Dietary Behaviors. This measure will be used to assess the various components of Social Cognitive Theory which are guiding the TeleSalud HE-PA/SB intervention.
Exercise Confidence Survey | Baseline, 4 months, 8 months
  Self-efficacy will be assessed by the Exercise Confidence Survey. This measure will be used to assess the various components of Social Cognitive Theory which are guiding the TeleSalud HE-PA/SB intervention.
Social Support and Eating Habits Survey | Baseline, 4 months, 8 months
  Social Support will be assessed by the Social Support and Exercise Survey and the Social Support and Eating Habits Survey. These measures will be used to assess the various components of Social Cognitive Theory which are guiding the TeleSalud HE-PA/SB intervention.
Social Support and Exercise Survey | Baseline, 4 months, 8 months
  Social Support will be assessed by the Social Support and Exercise Survey and the Social Support and Eating Habits Survey. These measures will be used to assess the various components of Social Cognitive Theory which are guiding the TeleSalud HE-PA/SB intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Sanchez-Johnsen, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States